CLINICAL TRIAL: NCT00526292
Title: Phase II Trial of HLA Haploidentical Natural Killer Cell Infusion for Treatment of Relapsed or Persistent Leukemia Following Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Chemotherapy and a Donor Natural Killer Cell Infusion in Treating Patients With Relapsed or Persistent Leukemia or Myelodysplastic Syndrome After a Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-035; FD-R-004128
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; blastic phase chronic myelogenous leukemia; previously treated myelodysplastic syndromes; childhood myelodysplastic syndromes; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; childhood chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Blast Crisis; Congenital Abnormalities | interventions — Cyclophosphamide; fludarabine

ARMS (1):
- natural killer (NK) cells with salvage chemotherapy (Experimental): This is a Phase II study, designed to determine the efficacy of natural killer (NK) cells isolated from HLA-haploidentical related donors when infused following a salvage chemotherapy regimen into patients who have relapsed or persistent leukemia following an allogeneic HLA-compatible HSCT and who are ineligible for a second HSCT.
  Interventions: Biological: natural killer cell therapy; Drug: cyclophosphamide; Drug: fludarabine

INTERVENTIONS:
Biological: natural killer cell therapy — The patient must be admitted by Day -8 to the Bone Marrow Transplant Service. On Day 0, patients will receive a single dose of allogeneic NK cells isolated from a HLA-haploidentical related donor and will be monitored for hematopoietic recovery.
Drug: cyclophosphamide — Day -6 cyclophosphamide 60mg/kg infused over 1 hour (dose adjusted for body weight) for 2 days
Drug: fludarabine — Day -5 fludarabine 25mg/m2 CIV for 5 days

SUMMARY:
The goal of this study is to see if there is a benefit to giving chemotherapy and then natural killer (NK) cells. The NK cells must come from a family member who shares half of the patients HLA proteins. NK cells are a type of white blood cell. They can recognize and kill abnormal cells in the body.

Patients whose blood cancer is not cured with a stem cell transplant do not have standard treatment options. Studies have shown that NK cells from a donor can be given safely and can be helpful in treating some blood diseases. These NK cells are collected from the patients donor and purified using a separation system called CliniMACS that has been used safely in previous studies and is used in this study with the approval of the Federal Food and Drug Administration. The researchers want to find out what effects the NK cells will have on blood cancer and bone marrow function and how to maximize its benefits in treating blood cancers. The researchers hope that giving chemotherapy and then NK cells will be a better treatment for the disease than the current available treatment options.

Funding Source - Food and Drug Administration/Office of Orphan Products Development

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the anti-leukemic efficacy of allogeneic HLA-haploidentical related natural killer (NK) cell infusion following a cytoreductive regimen with cyclophosphamide and fludarabine in patients with acute myeloid leukemia (AML), myelodysplastic syndromes (MDS), or blastic CML who have relapsed following allogeneic hematopoietic stem cell transplant, where efficacy is defined as the achievement of complete or partial remission at one year following NK cell infusion.

Secondary

* To assess treatment efficacy, as defined by achievement of complete or partial remission, at 3 and 6 months following HLA-haploidentical related NK cell infusion.
* To assess the effects of an HLA-haploidentical related NK cell infusion on the sustained engraftment and recovery of an HLA-matched stem cell allograft.
* To assess the risk of inducing graft-vs-host disease (GVHD) or altering its severity.
* To provide preliminary evidence that specific donor KIR-recipient HLA ligand combinations relating to missing self-MHC class I ligand or missing class I ligand are associated with higher NK alloreactivity and improved outcome.
* To monitor the extent and duration of NK cell donor chimerism.
* To monitor NK cell reconstitution through NK receptor cell surface phenotyping (CD94/NKG2A, ILT-2, KIR expression) and function (intracellular IFN-γ, cytotoxicity) on day 15, 30, 60, 100, and 200 following the NK infusion and to correlate with outcome.
* To correlate the magnitude of NK effect with disease and known survival risk factors (time from allogeneic HSCT to relapse; < 6 months vs > 6 months).

ELIGIBILITY:
Subject Inclusion Criteria:

Diagnosis and Status

* Patients with a pathologically confirmed diagnosis of relapsed or persistent resistant AML, MDS, or blastic CML following HSCT and who have been deemed ineligible for second HSCT after consideration of adequacy of their physical function, extent of disease, and prior treatment-related toxicities.

Eligible patients have evidence of disease with ≥5% bone marrow involvement detected by morphology or abnormal cytogenetics (by karyotype or FISH). Patients with molecular detection of markers characteristic of the patient's disease from two consecutive bone marrow biopsies are also eligible. Following diagnosis of relapsed disease, treatment to reduce leukemic burden is allowed prior to protocol therapy without the need for additional disease documentation prior to cyclophosphamide and fludarabine.

* Patients with extramedullary relapse are eligible except for those with CNS involvement.
* Patients must have received an allogeneic HSCT.
* Patient must not be pregnant and must be using adequate form of birth control.
* Patients must have a Karnofsky (adult) or Lansky (pediatric) Performance Status ≥ 60%.
* Hospitalization does not preclude enrollment, as long as the patient's performance status is ≥ 60% according to the KPS grading scale.
* Patients must have adequate physical function measured by :

Cardiac: asymptomatic and LVEF at rest must be > 50%. Hepatic: < 2x ULN ALT and < 1.5 total serum bilirubin, unless liver is involved with disease, there is congenital benign hyperbilirubinemia, or other reversible causes of hepatic abnormalities are documented.

Renal: serum creatinine <1.5 mg/dl or if serum creatinine is outside the normal range, then CrCl > 50 ml/min Pulmonary: Patient cannot be oxygen-dependent.

* Patients with documented GVHD are not excluded from this trial, but either must not have used systemic immunosuppression for two weeks, or during immunosuppression taper have documented two subtherapeutic levels at least one week apart. Immunosuppressive agents include but are not limited to systemic steroids, calcineurin inhibitors, MTOR-inhibitors, Budesonide, anti-thymocyte globulin. The maximal allowable dose of corticosteroids is the equivalent of 10 mg/day prednisone.
* Patients with grade I/II acute GVHD or limited chronic GVHD and receiving localized GVHD therapy (e.g. topical steroids) are not excluded from this trial.
* Patients having received previous adoptive cellular therapy such as donor lymphocyte infusion (DLI) are not excluded from this trial as long as their disease has been documented to progress within two months of receiving DLI or if the patient has not received DLI within two months of NK cell infusion.
* Patients who have received cytoreductive therapy following documentation of relapse and prior to enrollment are not excluded from this trial. The interval between standard reinduction chemotherapy and start of protocol chemotherapy should be a minimum of 2 weeks, and all induction chemotherapy-related toxicities should be documented to be completely resolved. For patients receiving nonintensive chemotherapies such as hydroxyurea or low-dose cytarabine, nonintensive chemotherapies should be discontinued upon initiation of protocol chemotherapy.
* Each patient must be willing to participate as a research subject and must sign an informed consent form. Parents or legal guardians of patients who are minors may sign the informed consent form
* Patients must have an eligible NK donor.
* There are no age restrictions to this protocol.

NK Cell Donor Eligibility

* Donor is blood-related and HLA-haploidentical to the recipient.
* Donor has undergone serologic testing for transmissible diseases as per blood banking guidelines for organ and tissue donors. Tests include but are not limited to: HepBsAg, HepBsAb, HepBcAb, HepC antibody, HIV, HTLV I and II, VZV, CMV and VDRL, and West Nile Virus . Donor must have normal negative test results for HIV, HTLV I and II, and West Nile Virus. Donor exposure to other viral pathogens will be discussed on a case-by-case basis by the Transplant team.
* Donor has a CXR and EKG performed.
* Donor must be able to undergo leukopheresis for total volume of 10-15 liters.
* Donor is not pregnant.
* Donor does not have concurrent malignancy or autoimmune disease.
* There is no age restriction for the donor.

Subject Exclusion Criteria:

* Patients on systemic immunosuppression with therapeutic drug levels. Patients whose immunosuppression is being actively tapered and have documentation of subtherapeutic drug levels one week apart are not excluded from enrollment. For patients receiving corticosteroids, the maximal allowable dose of corticosteroids is the equivalent of 10 mg/day prednisone.
* Patients with untreated or uncontrolled active infection. Infections that are controlled or being appropriately treated does not exclude a patient from enrollment.

NK Cell Donor Exclusion

* Donor has cardiac risk factors precluding ability to undergo leukopheresis.
* Donor has evidence of concurrent malignancy or autoimmune disease.
* Donor is pregnant.

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hsu, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Ann Alice Jakubowski, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HLA Haploidentical Natural Killer Cell Infusion: HLA Haploidentical Natural Killer Cell Infusion for Treatment of Relapsed or Persistent Leukemia
Period: Overall Study
Arm/Group | HLA Haploidentical Natural Killer Cell Infusion
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HLA Haploidentical Natural Killer Cell Infusion
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy as Defined by Complete or Partial Remission
Time Frame: 3 Months following treatment
Measure: Number; unit: participants
Arm/Group | HLA Haploidentical Natural Killer Cell Infusion
Number analyzed (Participants) | 6
participants
  Complete Remission | 1
  Progression of Disease (POD) | 5

ADVERSE EVENTS:
Arm/Group | HLA Haploidentical Natural Killer Cell Infusion
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HLA Haploidentical Natural Killer Cell Infusion (N=6)
Death not associated with CTCAE term-Disease progression NOS (General disorders) | 3
Febrile neutropenia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HLA Haploidentical Natural Killer Cell Infusion (N=6)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 6
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2
Platelets (Blood and lymphatic system disorders) | 6
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes